CLINICAL TRIAL: NCT06582459
Title: Efficacy and Safety of High-Flow Nasal Cannula Versus Noninvasive Ventilation for Pulmonary Arterial Hypertension-Associated Acute Respiratory Failure: a Retrospective Cohort Study Stratified by Right Ventricular Dysfunction Severity
Brief Title: Efficacy and Safety of High-Flow Nasal Cannula Versus Noninvasive Ventilation for Pulmonary Arterial Hypertension-Associated Acute Respiratory Failure
Acronym: HFCNV-PAH
Status: Active, not recruiting | Type: Observational
Sponsor: The First People's Hospital of Neijiang (Other)
Responsible Party: Principal Investigator, Ou Jiang, Director of Cancer Center, The First People's Hospital of Neijiang
Other Study IDs: 2021-lunshenpi-38
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension; Acute Respiratory Failure; High-flow Nasal Cannula; Noninvasive Ventilation
Keywords: Pulmonary hypertension, Acute respiratory failure, High-flow nasal cannula, Noninva-sive ventilation, Right ventricular dysfunction
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HFNC treatment: HFNC therapy. The initial flow rate of 50-60 L/min was subsequently adjusted to maintain an oxygen saturation (SpO2) ≥92%. The FiO2 was titrated to maintain the PaO2 between 60 and 80 mmHg.
  Interventions: Device: HFNC treatment
- NIV treatment: A Mindray SV300 ventilator (Mindray Medical International Limited, Shenzhen, China) was used to deliver NIV via an oronasal mask. The initial inspiratory positive airway pressure (IPAP) was 12-15 cmH2O and adjusted later to achieve a tidal volume of 6-8 mL/kg of predicted body weight and a respiratory rate of <30 breaths/min. The expiratory positive airway pressure (EPAP) was established at 5-8 cmH2O. Additional-ly, FiO2 was titrated to maintain a PaO2 between 60 and 80 mmHg.
  Interventions: Device: NIV treatment

INTERVENTIONS:
Device: HFNC treatment — HFNC treatment HFNC therapy. The initial flow rate of 50-60 L/min was subsequently adjusted to maintain an oxygen saturation (SpO2) ≥92%. The FiO2 was titrated to maintain the PaO2 between 60 and 80 mmHg.
  Groups: HFNC treatment
Device: NIV treatment — NIV treatment A Mindray SV300 ventilator (Mindray Medical International Limited, Shenzhen, China) was used to deliver NIV via an oronasal mask. The initial inspiratory positive airway pressure (IPAP) was 12-15 cmH2O and adjusted later to achieve a tidal volume of 6-8 mL/kg of predicted body weight and a respiratory rate of <30 breaths/min. The expiratory positive airway pressure (EPAP) was established at 5-8 cmH2O. Additional-ly, FiO2 was titrated to maintain a PaO2 between 60 and 80 mmHg.
  Groups: NIV treatment

SUMMARY:
This is a single center, retrospective, propensity score matching cohort study that explores the efficacy and safety of high flow nasal cannula and non-invasive ventilation in the treatment of acute respiratory failure associated with pulmonary arterial hypertension, stratified by the severity of right ventricular dysfunction.

The study will compare two groups: high flow nasal cannula (HFNC) and non-invasive ventilation (NIV).

Main objective: heart function parameters (e.g. TAPSE and RVSP) Secondary objectives: respiratory support success rate (defined as the avoidance of endotracheal introduction or death duration hospitalization), respiratory support duration, length of intensive care unit (ICU) stay, length of hospital stay, and in-hospital mortality.

This study addresses whether NIV or HFNC should be prioritized for the treatment of acute respiratory failure associated with pulmonary arterial hypertension in patients with severe right ventricular dysfunction who require high flow nasal cannula and non-invasive ventilation.

This study is of great significance as it is based on a patient stratification method of right ventricular dysfunction severity to evaluate the effectiveness of HFNC treatment and NIV in PH related ARF patients.

DETAILED DESCRIPTION:
Study Title: Efficiency and Safety of High Flow Nassal Cannula Versus Noninvasive Ventilation for Pulsary Arterial Hypertension Associated Acute Respiratory Failure: A Retrospective Cohort Study Stratified by Right Ventricular Dysfunction Severity Background: Patients with pulmonary hypertension (PH) typically have high morbidity and mortality when they develop acute respiratory failure (ARF) The best method of respiratory support considering the severity of right ventricular (RV) dysfunction is still uncertain.

Main objective: heart function parameters (e.g. TAPSE and RVSP) Secondary objectives: respiratory support success rate (defined as the avoidance of endotracheal introduction or death duration hospitalization), respiratory support duration, length of intensive care unit (ICU) stay, length of hospital stay, and in-hospital mortality.

Research Design: This is a single center, retrospective, propensity score matching cohort study.

The study will compare two groups: high flow nasal cannula (HFNC) and non-invasive ventilation (NIV).

Significance: This study aims to address whether NIV or HFNC should be prioritized for the treatment of acute respiratory failure associated with pulmonary arterial hypertension in patients with severe right ventricular dysfunction who require high flow nasal cannula and non-invasive ventilation.

Innovation: A patient stratification method based on the severity of right ventricular dysfunction to evaluate the effectiveness of HFNC treatment and NIV in PH related ARF patients.

Expected outcome: HFNC treatment is equally effective as NIV in treating mild to moderate right ventricular dysfunction; NIV may be more beneficial for critically ill patients. Assist PH patients with ARF in choosing between HFNC treatment and NIV.

Conclusion: Our study provides new insights into the comparative performance of HFNC therapy and NIV in patients with PH combined with ARF.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients aged ≥ 18 years old；
* Patients diagnosed with PH based on right ventricular systolic pressure (RVSP)>50 mmHg on echocardiography or right heart catheterization (resting mean pulmonary artery pressure ≥ 25 mmHg)；
* And patients who require HFNC or NIV respiratory support after ACRF (defined as acute deterioration of respiratory function in patients with chronic respiratory diseases, resulting in PaO2<60 mmHg, PaO2/FiO2 ratio<300 mmHg, or respiratory rate>30 breaths per minute in indoor air).

Exclusion Criteria:

* The exclusion criteria were patients with acute coronary syndrome, acute myocardial infarction, severe arrhythmias, severe cerebrovascular or neurological diseases, and severe hepatic or renal dysfunction;
* those who were receiving endotracheal intubation or NIV within 24 h of admission;
* patients who were not intubated;
* those who were receiving palliative care;
* immunocompromised patients;
* patients with incomplete data or who were lost to follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Inclusion criteria are patients aged ≥ 18 years old；
  2. Patients diagnosed with PH based on right ventricular systolic pressure (RVSP)>50 mmHg on echocardiography or right heart catheterization (resting mean pulmonary artery pressure ≥ 25 mmHg)；
  3. And patients who require HFNC or NIV respiratory support after ACRF (defined as acute deterioration of respiratory function in patients with chronic respiratory diseases, resulting in PaO2<60 mmHg, PaO2/FiO2 ratio<300 mmHg, or respiratory rate>30 breaths per minute in indoor air).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
heart function parameters | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  (e.g., TAPSE and RVSP) from baseline to 24 h after respiratory support initiation.

SECONDARY OUTCOMES:
respiratory support success rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  defined as the avoidance of endotracheal intubation or death during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Neijiang City, Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Background] Hoeper MM, Humbert M, Souza R, Idrees M, Kawut SM, Sliwa-Hahnle K, Jing ZC, Gibbs JS. A global view of pulmonary hypertension. Lancet Respir Med. 2016 Apr;4(4):306-22. doi: 10.1016/S2213-2600(15)00543-3. Epub 2016 Mar 12. PMID 26975810
- [Background] Campo A, Mathai SC, Le Pavec J, Zaiman AL, Hummers LK, Boyce D, Housten T, Lechtzin N, Chami H, Girgis RE, Hassoun PM. Outcomes of hospitalisation for right heart failure in pulmonary arterial hypertension. Eur Respir J. 2011 Aug;38(2):359-67. doi: 10.1183/09031936.00148310. Epub 2011 Feb 10. PMID 21310884
- [Background] Sztrymf B, Souza R, Bertoletti L, Jais X, Sitbon O, Price LC, Simonneau G, Humbert M. Prognostic factors of acute heart failure in patients with pulmonary arterial hypertension. Eur Respir J. 2010 Jun;35(6):1286-93. doi: 10.1183/09031936.00070209. Epub 2009 Nov 6. PMID 19897557
- [Background] Kurzyna M, Zylkowska J, Fijalkowska A, Florczyk M, Wieteska M, Kacprzak A, Burakowski J, Szturmowicz M, Wawrzynska L, Torbicki A. Characteristics and prognosis of patients with decompensated right ventricular failure during the course of pulmonary hypertension. Kardiol Pol. 2008 Oct;66(10):1033-9; discussion 1040-1. PMID 19006024
- [Background] Atwood CW Jr, McCrory D, Garcia JG, Abman SH, Ahearn GS; American College of Chest Physicians. Pulmonary artery hypertension and sleep-disordered breathing: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):72S-77S. doi: 10.1378/chest.126.1_suppl.72S. PMID 15249496
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Ferreyro BL, Angriman F, Munshi L, Del Sorbo L, Ferguson ND, Rochwerg B, Ryu MJ, Saskin R, Wunsch H, da Costa BR, Scales DC. Association of Noninvasive Oxygenation Strategies With All-Cause Mortality in Adults With Acute Hypoxemic Respiratory Failure: A Systematic Review and Meta-analysis. JAMA. 2020 Jul 7;324(1):57-67. doi: 10.1001/jama.2020.9524. PMID 32496521
- [Derived] Yu L, Chen X, Wang X, Cui R. Efficacy and safety of high-flow nasal cannula versus noninvasive ventilation for pulmonary arterial hypertension-associated acute respiratory failure: A retrospective cohort study stratified by the severity of right ventricular dysfunction. Medicine (Baltimore). 2025 Jul 4;104(27):e43185. doi: 10.1097/MD.0000000000043185. PMID 40629562